CLINICAL TRIAL: NCT05862844
Title: PROMIS WOMAN Education Program : ImProving ceRvical Cancer preventiOn Methods Among Muslim AmerIcans WOMEN
Brief Title: Promise Women Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Dignan, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Virginia Commonwealth University (Other)
Responsible Party: Sponsor-Investigator, Mark Dignan, PhD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HM20024502_VCU; 3P30CA177558-10S1 (NIH)
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Human Papilloma Virus; Cervical Cancer
Keywords: screening; vaccination; Muslim American women; prevention; Health disparities; Acceptability and feasibility.; Behavioral intervention; Religious adaptation
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: In this study, the investigators will conduct a single-arm pilot trial using a pre-and post-test survey design to evaluate the effectiveness of a religiously tailored and culturally appropriate intervention program for promoting cervical cancer prevention among Muslim American women. 20 eligible participants who have not previously participated in our studies will be recruited. Before the intervention, participants will complete a pre-intervention survey to assess their knowledge and acceptance of cervical cancer prevention. Following the intervention, participants will undergo the post-intervention survey to measure any changes in their knowledge and acceptance levels. By utilizing this survey-based approach, the investigators aim to gather valuable data on the impact of the intervention and determine its potential effectiveness in improving participants' understanding and engagement with cervical cancer prevention activities.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The single-arm trial with a pre- and post-test design (Experimental): The Intervention Arm in the Promise Women Project evaluates a specific educational intervention program for Muslim women to promote cervical cancer prevention. It involves a one-time, 90-minute culturally and religiously tailored educational session with 20 participants. The session covers perceived risks of Human Papilloma Virus (HPV) infection, cervical cancer, and benefits of early screening and vaccination. Pre- and post-intervention surveys measure changes in participants' knowledge. This experimental arm assesses the intervention's effects on knowledge and acceptance of cervical cancer prevention.
  Interventions: Behavioral: Promise women project (Promote Cervical Cancer Prevention Methods Among Muslim Women in Virginia )

INTERVENTIONS:
Behavioral: Promise women project (Promote Cervical Cancer Prevention Methods Among Muslim Women in Virginia ) — The Intervention Arm involves a 90-minute educational session tailored to Muslim women. They will learn about HPV infection risks, cervical cancer risks, and benefits of early screening and HPV vaccination. Discussions cover transmission, consequences, risk factors (behaviors, infections, family history), and importance of early detection. The session provides information on screening methods, check-ups, and HPV vaccine safety. Participants actively engage in discussions, ask questions, and share thoughts. The session empowers women with knowledge to make informed decisions about their health, promoting cervical cancer prevention.
  Other Names: Culturally tailored educational session on cervical cancer prevention

SUMMARY:
The goal of this study is to develop and test an intervention program to improve cervical cancer prevention among Muslim American women. The main questions the investigators aim to answer are:

* Will the religiously tailored and culturally appropriate intervention program improve participants' knowledge and acceptance of cervical cancer prevention?
* Is the intervention program feasible to conduct and acceptable to participants?

Participants will be asked to:

* Attend focus group sessions to provide input on the development of educational materials.
* Complete pre- and post-intervention surveys to measure changes in knowledge and acceptance of cervical cancer prevention.
* Engage in the intervention program, which includes education and experiential practice/communication skills training.
* Provide feedback through satisfaction surveys. Researchers will compare participant outcomes before and after the intervention to assess its effectiveness. Additionally, the program's feasibility and acceptability will be evaluated based on enrollment rates, successful implementation, participant engagement, retention, and satisfaction.

DETAILED DESCRIPTION:
This project involves creating special educational materials for Muslim women to learn about cervical cancer prevention. The investigators will engage in discussions with 10 Muslim women during dedicated group sessions to ensure the suitability of the materials. They will also seek input from Muslim religious leaders. Subsequently, they will conduct surveys before and after the program to assess the effectiveness of the materials in facilitating women's learning and comprehension of cervical cancer prevention. To determine its efficacy and acceptability, the investigators will implement the program with an additional 20 women and gather their feedback. The goal of this project is to promote the health and well-being of Muslim women by providing them with culturally and religiously sensitive information regarding cervical cancer prevention.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Female Muslim individuals above 18 years old.
* Able to speak and understand English.
* Have not had a hysterectomy.
* Have not had a cervical cancer diagnosis.
* Willing to participate in the educational program and undergo cervical cancer screening.
* Physically well, able to give consent form.

Exclusion Criteria:

* Under age 18
* Not Muslim
* Unable to provide consent
* Participated in a pilot study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa L Sheppard, PhD, Study Director — Virginia Commonwealth University; Mark B Dignan, PhD, MPH, Study Director — University of Kentucky
Locations (4):
- United States (4):
  - the Islamic center of Hampton, Hampton, Virginia
  - the Peninsula Islamic Community Center, Hampton, Virginia
  - Islamic center of Henrico-Alfalah, Henrico, Virginia
  - the Islamic center of Richmond, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The Single-arm Trial With a Pre- and Post-test Design
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | The Single-arm Trial With a Pre- and Post-test Design
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (14.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 7
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Who Undergo Cervical Cancer Screening.
Description: measured by tracking the number of women who schedule and attend
Time Frame: Baseline and Post Intervention (up to 1 week)
Measure: Count of Participants; unit: Participants
Arm/Group | The Single-arm Trial With a Pre- and Post-test Design
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Number of Women Enrolled
Description: Test the intervention program's feasibility as evidenced by meeting enrollment targets
Time Frame: Baseline and Post Intervention (up to 1 week)
Measure: Count of Participants; unit: Participants
Arm/Group | The Single-arm Trial With a Pre- and Post-test Design
Number analyzed (Participants) | 20
Participants | 20

3. Other Pre Specified Outcome: Number of Women That Attend the Education Session
Description: Test the intervention program's acceptability as evidenced by session attendance
Time Frame: Baseline and Post Intervention (up to 1 week)
Measure: Count of Participants; unit: Participants
Arm/Group | The Single-arm Trial With a Pre- and Post-test Design
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: Baseline and Post Intervention (up to 1 week)
Arm/Group | The Single-arm Trial With a Pre- and Post-test Design
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT05862844/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT05862844/ICF_000.pdf